CLINICAL TRIAL: NCT05618834
Title: Optimizing Daily Care Interactions Between Staff and Assisted Living Residents With Alzheimer's Disease and Related Dementias
Brief Title: Promoting Positive Care Interactions (PPCI) in Assisted Living
Acronym: PPCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Anju Paudel, PhD, MGS, RN, Assistant Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00021256
Record Dates: First submitted 2022-10-31; First posted 2022-11-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease and Related Dementias
Keywords: Dementia; Care Interactions; Communication; Assisted Living; Long-Term Care
MeSH Terms: conditions — Alzheimer Disease; Dementia; Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPCI Arm (Experimental): The ALF/PCH assigned as treatments will receive the four steps of PPCI including, stakeholder engagement and facility goal development, environment and policy assessment, staff education, and ongoing mentorship/motivation and support over a period of six-months by a research nurse facilitator (RNF), a registered nurse (RN) with prior experience in long-term care. The RNF will work with an identified internal/facility champion monthly to implement the four steps of PPCI.
  Interventions: Behavioral: Promoting Positive Care Interactions (PPCI)
- PPCI-Staff Education Only Arm (Active Comparator): The ALF/PCH assigned as controls will receive PPCI-staff education only (EO). The EO will include a 30-45 min in-service session and monthly f/u visits for booster education. The education content and process will be the same as outlined in Step 3 of the PPCI for treatment sites.
  Interventions: Behavioral: PPCI-Staff Education Only (EO)

INTERVENTIONS:
Behavioral: Promoting Positive Care Interactions (PPCI) — The PPCI consists of four steps: (1) stakeholder engagement in developing facility specific goals; (2) environment and policy assessments; (3) flexible staff education; and (4) ongoing mentorship, motivation, and support (in-person visits and text messages) for staff to optimize care interactions.
  A research nurse facilitator (RNF), a registered nurse (RN) with prior experience in long-term care will work with an identified internal champion monthly to implement the four steps of PPCI. The PPCI intervention comprehensively focuses on intrapersonal, interpersonal, organizational, and environmental/policy factors to bring together evidence and key stakeholders to optimize daily care interactions in assisted living.
  Arms: PPCI Arm
Behavioral: PPCI-Staff Education Only (EO) — The EO will include a 30-45 min in-service session and monthly f/u visits for booster education. The education content and process will be the same as outlined in Step 3 of the PPCI for treatment sites.
  Arms: PPCI-Staff Education Only Arm

SUMMARY:
The overall aim of this study is to pilot test Promoting Positive Care Interactions (PPCI) with the goal of establishing a feasible and culturally responsive approach to optimize care interactions between staff (nursing, activity, housekeeping, and dining service staff) and residents with ADRD in assisted living facilities (ALFs), and further improve select resident, staff, and facility outcomes. PPCI is a non- pharmacological four-step approach consisting of (1) stakeholder engagement in developing facility specific goals; (2) environment and policy assessments; (3) flexible staff education; and (4) ongoing mentorship, motivation, and support (in-person visits and text messages) for staff to optimize care interactions.

DETAILED DESCRIPTION:
Nearly one million individuals living in 28,900 assisted living facilities (ALFs) in the U.S. participate in daily care interactions, defined as any verbal or nonverbal exchange between staff and residents during physical and social care activities. While there are positive care interactions, poor care interactions also persist with prevalence as high as 25% in long-term care including ALFs. Individuals with Alzheimer's disease and related dementias (ADRD) are especially at risk for poor care interactions due to ineffective staff approaches such as negative touching (e.g., quickly removing clothes to bathe a resident), being overprotective (e.g., restricting activity for safety concerns), and lack of verbal or non-verbal contact during care. Persistent poor care interactions can negatively affect both residents and staff. Thus, there is a need to replace poor care interactions with positive care interactions, now more than ever given the worsening staff retention related to COVID-19 pandemic, and constant need to train new employees.

Positive care interaction refers to care interactions where staff use positive approaches such as honoring resident's abilities and preferences, recognizing resident's responses/non-verbal cues, acknowledging resident's effort, providing role modeling and verbal cues, managing self-responses, and using a calm respectful approach for appropriate delivery of care. It has been long known that use of positive approaches benefits both residents (e.g., less behavioral distress) and staff (e.g., greater competence in care). Yet, poor interactions continue in ALFs due to interlocking barriers associated with residents' ADRD-related communication and other difficulties and behaviors of distress (e.g., agitation), as well as staff's knowledge and training deficits in ADRD care; ALFs have fewer licensing and training mandates for staff. Lack of cultural concordance can also contribute to poor interactions. The ALF staff, often younger (mean age=38.3 yrs.) females (83.8%) with almost half representing racial minorities (47.6%) care for largely non-Hispanic white (81.4%) resident population >=65 years (93.4%). Additionally, there are systemic barriers including limited organizational engagement in implementing and sustaining these approaches, lack of environmental infrastructure (e.g., controlled noise and availability of augmentative devices such as pocket talker) and policies (e.g., consistent assignments) to support positive care interactions, and lack of adequate mentoring and support for staff. It is crucial to address these issues and barriers and train ALF staff on positive care interactions, particularly since prior work has targeted nursing homes and focused on social interactions or verbal communication.

Therefore, this study proposes Promoting Positive Care Interactions (PPCI), a four-step approach, based on Social Ecological Model (SEM) and Social Cognitive Theory (SCT), to optimize daily care interactions between staff and residents with ADRD in ALFs. The four steps include: 1) stakeholder engagement in developing facility specific goals; (2) environment and policy assessments; (3) flexible staff education; and (4) ongoing mentorship, motivation, and support (in-person visits and text messages) for staff to optimize care interactions. These four steps are based on prior work implementing function & behavior focused intervention studies but have never been used in a care interaction-focused intervention nor been tested for cultural responsiveness. This study will follow a cluster randomized trial in a sample of 60 residents and 60 staff in four ALFs in central PA (approx. 15 residents, 15 staff/ALF) who agree and consent to participate in this study. The treatment group will receive all four steps of PPCI while the control arm will receive education only.

ELIGIBILITY:
Inclusion Criteria:

Assisted Living Facility (ALF) will be included in the study if they:

1. have at least 20 or more beds
2. are able to identify a facility champion, and
3. express a willingness to actively partner in an initiative to change practice at their institution

Staff will be included in the study if they:

1. are able to communicate in English, and
2. work at least 16 hours a week at the facility at the time of recruitment in nursing, activities, housekeeping, or dining service roles

Residents will be included in the study if they:

1. are 65 years old or greater
2. are living at the facility at the time of recruitment, and
3. have a diagnosis of ADRD and Saint Louis University Mental Status Exam (SLUMS) score of 20 or less (high school education)/ 19 or less (less than high school education) suggesting ADRD

Exclusion Criteria:

Assisted Living Facility (ALF) will be excluded from the study if they:

1. have less than 20 beds
2. are unable to identify a facility champion, and
3. do not express a willingness to actively partner in an initiative to change practice at their institution

Staff will be included in the study if they:

1. are unable to communicate in English, and
2. work less than16 hours a week at the facility at the time of recruitment in nursing, activities, housekeeping, or dining service roles

Residents will be included in the study if they:

1. are less than 65 years old
2. are not living at the facility at the time of recruitment, and
3. do not have a diagnosis of ADRD and Saint Louis University Mental Status Exam (SLUMS) score of 20 or less (high school education)/ 19 or less (less than high school education) suggesting ADRD

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The degree to which the intervention can be implemented as intended assessed by Feasibility of Intervention Measure (FIM) Questionnaire | six-months post intervention
  4 items answered on a 5-point ordinal scale ranging from 'completely disagree' to 'completely agree'; range = 4 to 20 and higher scores are better
The degree to which the intervention is acceptable assessed by Acceptability of Intervention Measure (AIM) Questionnaire | six-months post intervention
  4 items answered on a 5-point ordinal scale ranging from 'completely disagree' to 'completely agree'; range = 4 to 20 and higher scores are better

SECONDARY OUTCOMES:
Well-being assessed by Quality of Life in Late-stage Dementia (QUALID) Scale | baseline and 6 months
  11 items on a 5-point scale, range = 11 to 55 and higher scores are better
Level of agitation assessed by Cohen-Mansfield Agitation Inventory (CMAI-short form) | baseline and 6 months
  14 items answered on a 5-point scale, range = 14 to 70 and lower scores are better
Frequency and intensity of resistive behaviors assessed by Resistiveness to Care (RTC) Scale | baseline and 6 months
  13 items answered on a 3-point scale for intensity and a number provided for frequency, range = 13 to 39 for intensity and lower scores are better
Knowledge of person-centered behavioral approaches for managing behavioral symptoms of distress assessed by Knowledge of Person-Centered Behavioral Approaches for BPSD | baseline and 6 months
  10 items with four responses (1 correct, 3 distracters), range = 0 to 10 and higher scores are better
Perceived competence in dementia care assessed by Sense of Competence in Dementia Care Staff (SCIDS) | baseline and 6 months
  17 items on a 4-point scale, range = 17 to 68 and higher scores are better
Level of stress assessed by Health Professions Stress Inventory (HPSI) | baseline and 6 months
  12 items on a 5-point scale, range = 0 to 48 and lower scores are better
Staff-resident relationship quality assessed by Positive Affect Index (PAI) | baseline and 6 months
  5 items on a 6-point scale, range = 5 to 30 and higher scores are better
Staff-resident care interactions assessed by Quality of Care Interactions Schedule (QuIS) | baseline and 6 months
  5 items answered on a 3-point scale, range = 0 to 7 and higher scores are better
Provision of facility policies pertaining to promoting positive care interactions (PPCI) assessed by Assessment of Policies for PPCI | baseline and 6 months
  24 items answered as yes (1) or no (0), range = 0 to 24 and higher scores are better
Provision of facility environment pertaining to promoting positive care interactions (PPCI) assessed by Assessment of Environment for PPCI | baseline and 6 months
  23 items answered as yes (1) or no (0), range = 0 to 23 and higher scores are better

OTHER OUTCOMES:
Cultural responsiveness assessed by a questionaire based on the ecological model (EM) domains: language, persons, metaphors, goals, content, concepts, methods, & context of PPCI | six-months post intervention
  12 interview questions

CONTACTS AND LOCATIONS:
Overall Officials: Anju Paudel, Assistant Professor, Principal Investigator — Penn State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No